CLINICAL TRIAL: NCT03458195
Title: Ileal Crohn's Disease and Post-operative Outcome: Prospective Cohort Study of the REMIND Group
Acronym: POP-REMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Principal Investigator, Madeleine Bezault, Pr Matthieu Allez, Saint-Louis Hospital, Paris, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: POP STUDY - REMIND
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Crohn Disease
Keywords: ileo-caecal resection; post-operative recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients aged 18 or more, for whom Crohn's disease diagnosis is confirmed and ileum or ileocecal Crohn's disease require surgical resection. in addition to usual practice, a bio-banking (blood samples, biopsies and surgical specimens) is collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crohn's disease patients (Experimental): Patients aged 18 or more, for whom Crohn's disease diagnosis is confirmed and ileum or ileocecal Crohn's disease require surgical resection. in addition to usual practice, a bio-banking (blood samples, biopsies and surgical specimens) is collected.
  Interventions: Other: bio-banking collection

INTERVENTIONS:
Other: bio-banking collection — blood samples, biopsies, and surgical specimen collected in addition to usual practice

SUMMARY:
Crohn's disease (CD), a chronic inflammatory process in intestinal segments leads to tissue damage. More than two thirds of CD patients need intestinal resection. Symptomatic clinical recurrence occurs in 60% by 10 years. The principal factors affecting postoperative recurrence are active smoking, penetrating disease, perianal lesions history, prior intestinal resection, small bowel resection extent, and prophylaxis treatment absence.

Ileocolonoscopy within one year of surgery can predict clinical recurrence risk.

Different therapies are proposed after surgery, to prevent post-operative recurrence : Thiopurines, 6-mercaptopurine (positive for clinical and endoscopic postoperative recurrence prevention), Anti-tumour necrosis factor therapy (anti-TNF), the most effective therapy.

Intestinal microbiota acts as a central factor in the CD pathogenesis, and fecal stream role is clearly shown. Various changes in luminal flora with a possible link to local inflammation was also demonstrated. Bacteria associated with postoperative recurrence could be more pathogenic as adherent invasive E coli (AIEC), which could be a pathogen in CD through several mechanisms including increased mucosal colonization, adherence, replication and induction of TNF secretion. Alternatively, postoperative CD recurrence could be linked to a protective commensal species lack, such as Faecalibacterium prausnitzii.

Microscopic inflammation occurs as early as 8 days after anastomosis in the neoterminal ileum mucosa. IL6, IL10 and TGFb levels, measured in neoterminal ileum early after surgery are associated with different rates of postoperative recurrence. It suggests cytokines implication in postoperative recurrence. T cells are major players in the intestinal immune response. The presence at time of surgery and persistence of disease inducing T cell clonal expansions could play an important role in post-operative recurrence.

The main objective is to define a classification of ileal Crohn's Disease based on data integration on a large cohort of patients.

DETAILED DESCRIPTION:
Crohn's Disease is a major health issue with a complex etiology and despite available medical treatment, patients endure poor quality of life. The disease 's characterization on a molecular level will allow for a better management of patients treatment. To do so, the strategy is to integrate precise prospective clinical records with extensive biological data in a large cohort of patients.

All the clinical centers, participating to the study, include patients, with a tight collaboration between Gastroenterology and Surgery departments. Demographics and clinical parameters are collected in an eCRF.

Inclusion of patients is performed, before a scheduled ileocecal resection or ileal resection, and after eligibility criteria checking, and consent form signature. During surgery, several samples are collected : blood samples, mucosal biopsies, and surgical specimens. As usual practice, post-operative treatment will be prescribed at investigator's discretion, with help of a pre-established algorithm. Then, an endoscopic exam is scheduled, at least 6 months after surgery, or at least 6 months after intestine continuity restoration, in case of temporary stoma. Several samples are also collected during this exam (blood, ileal and colon biopsies).

At the same time as these 2 visits, clinical data regarding medical history, CD history, surgical history, treatments history, post-operative treatment if prescribed, treatments history between surgery and colonoscopy 6 months later, endoscopic score. Clinical data are also collected 18 months after surgery during a scheduled visit organized as usual practice, for long-term study : Clinical relapse, surgical recurrence, change in the therapy, hospitalizations and complications A patient has achieved the study after the endoscopic exam.

Several studies will be performed along the cohort setting-up:

* Transcriptomic analyses of mucosal tissues:
* Identification of a molecular signature predictive of post-operative recurrence
* Molecular classification of ileal Crohn's Disease
* Study of the mucosa-associated microbiota
* Study of association of AIEC
* Study of anti-TNF efficacy in post-operative recurrence prevention
* Study of new biologics in the treatment of post-operative recurrence All the biologic samples are stored on sites at -80°C, or at room temperature depending on the samples : Samples collected in Formol tubes, are sent immediatly, at room temperature, to the central pathology department in Beaujon Hospital, Paris. All the other samples, stored at -80°C, are sent to a central department, the Bio-Bank of Pasteur Hospital, Nice (every 3 months).

Samples analyses are performed by dedicated research centers: DNA, and RNA extraction for transcriptome analysis, Micobiota analysis, Lipids analysis, AIEC analysis :

Histological analyzes: Analyzis of the structure and inflammatory status of intestinal tissue of patients of the cohort, particularly at the ileal limit of the surgical specimens.

Molecular Biology: Whole genome expression analyses are performed using microarray and followed by Gene Ontology and clustering analyses.

Microbiology:

Adherent Invasive E.Coli (AIEC): The search for AIEC bacteria is carried out by culturing and investigating the characteristics of adhesion, invasion in Int-407 cells, and survival within THP-1 macrophages.

Microbiota: Bacterial composition of the ileal mucosa associated microbiota is analyzed at time of surgery using 16S (MiSeq, Illumina) sequencing. The obtained sequences are analyzed using the Qiime pipeline to assess composition, alpha and beta diversity.

Immunology:

Phenotype of mucosal and peripheral immune cells: Immune cells are extracted from blood and fresh mucosal tissues. The phenotype of these cells is analyzed by cytometry.

T cell repertoire: T cell receptor analysis on DNA extracted from biopsies is performed by next generation sequencing (Adaptive Biotechnology Inc., Seattle, Washington, USA). It is hypothesized that the persistence of these clonal expansions could be linked to the presence of specific microbial antigens.

Data Integration: The aim is to predict post-operative recurrence at M6. Integration of all datasets will explore the ability to predict post-operative recurrence. This will also allow to establish a molecular classification of CD, similar to what is already available in the oncology field. It will also be tried to find regulatory genes of the intestinal mucosa ("hubs"), using causal models (Bayesian networks) and co-expression networks (WCGNA). These findings could help drive potential innovative therapy for the treatment of CD.

The comparative analysis of the mucosa-associated transcriptome and microbiome will be performed. This could allow to elucidate the relations between bacteria and the intestinal mucosa, and to uncover pathways implicated in the bacteria-mucosa dialog. The correlations between certain groups of bacteria and the activation of a number of genes will be looked at. And genes known to play a role in the interaction between the microbiome and the mucosa will be specifically studied (MUC, DEF, REG, NOD2, …).

Lastly, once the patient genotypes will be available, an analysis of the genome together with the transcriptome and the relationship between genotype, transcriptome, and microbiome will be performed.

This analysis should help to robustly identify major pathways involved in intestinal inflammation, study the role played by genetics, and the impact on the gut microbiome. And finally to correlate these results with carefully curated clinical data: relapse/remission, post-operative recurrence, efficacy of post-operative therapies (anti TNF agents, ustekinumab).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities
* A diagnosis of CD, based on clinical, radiologic, endoscopic, or histological evidence.
* Men and women ≥18 years of age
* Required surgical intervention consisting in an ileocecal resection

Exclusion Criteria:

* Previous history of dysplasia or cancer in the ileum or colon
* Unwillingness or inability to follow the procedures outlined in the protocol
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Estimated)
Dates: Start 2009-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ileal Crohn's disease classification | surgery time, Time 0
  Ileal Crohn's disease classification will be performed using data integration (taking into account clinical data, immunological, genetic, microbiota, transcriptome data). A molecular classification will be possible due to this data integration analysis
Postoperative recurrence study | 6 months after surgery
  Rates of endoscopic recurrence as defined by a Rutgeerts score ≥ 1 in patients will be evaluated at the endoscopic exam
Study of Treatments efficacy to prevent recurrence | 6 months after surgery time
  During a clinical visit, scheduled as usual practice 6 months after surgery, clinical data will be collected : treatment modification or optimization, recurrence occurrence. If treament modification or optimization is needed (clinical symptoms or endoscopic recurrence), or complication occurs (abcess, occlusive syndrom, new surgery), patient will be considered as suffering a long-term relapse
Identification of biomarkers which could predict postoperative recurrence and response to treatments | surgery time, Time 0
  Identification of biomarkers taking into account clinical data, immunological, genetic, microbiota, transcriptome data

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu ALLEZ, Pr, Principal Investigator — Remind
Locations (17):
- SART Tilman Hospital, Liège, Belgium
- France (16):
  - Amiens Hospital, Amiens
  - Haut-levêque Hospital, Bordeaux
  - Clermont-Ferrand Hospital, Clermont-Ferrand
  - Beaujon Hospital, Clichy
  - Henri Mondor Hospital, Créteil
  - Kremlin-Bicêtre Hospital, Le Kremlin-Bicêtre
  - Lille Hospital, Lille
  - Hôpital Nord, CHU Marseille, Marseille
  - Montpellier Hospital, Montpellier
  - Brabois Hospital, Nancy
  - Nantes Hospital, Nantes
  - Archet 2 Hospital, Nice
  - Saint Louis Hospital, Paris
  - Saint Antoine Hospital, Paris
  - South Lyon Hospital, Pierre-Bénite
  - Strasbourg Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sokol H, Brot L, Stefanescu C, Auzolle C, Barnich N, Buisson A, Fumery M, Pariente B, Le Bourhis L, Treton X, Nancey S, Allez M, Seksik P; REMIND Study Group Investigators. Prominence of ileal mucosa-associated microbiota to predict postoperative endoscopic recurrence in Crohn's disease. Gut. 2020 Mar;69(3):462-472. doi: 10.1136/gutjnl-2019-318719. Epub 2019 May 29. PMID 31142586
- [Result] Auzolle C, Nancey S, Tran-Minh ML, Buisson A, Pariente B, Stefanescu C, Fumery M, Marteau P, Treton X, Hammoudi N; REMIND Study Group Investigators; Jouven X, Seksik P, Allez M. Male gender, active smoking and previous intestinal resection are risk factors for post-operative endoscopic recurrence in Crohn's disease: results from a prospective cohort study. Aliment Pharmacol Ther. 2018 Nov;48(9):924-932. doi: 10.1111/apt.14944. Epub 2018 Aug 20. PMID 30126030
- [Result] Allez M, Auzolle C, Le Bourhis L, Seksik P. Editorial: predicting recurrence of Crohn's disease after surgical resection-Close to a crystal ball. Authors' reply. Aliment Pharmacol Ther. 2018 Nov;48(10):1157-1158. doi: 10.1111/apt.14998. No abstract available. PMID 30375683
- [Result] Le Baut G, O'Brien C, Pavli P, Roy M, Seksik P, Treton X, Nancey S, Barnich N, Bezault M, Auzolle C, Cazals-Hatem D, Viala J, Allez M; REMIND GROUP; Hugot JP, Dumay A. Prevalence of Yersinia Species in the Ileum of Crohn's Disease Patients and Controls. Front Cell Infect Microbiol. 2018 Sep 21;8:336. doi: 10.3389/fcimb.2018.00336. eCollection 2018. PMID 30298122
- [Result] Allez M, Auzolle C, Ngollo M, Bottois H, Chardiny V, Corraliza AM, Salas A, Perez K, Stefanescu C, Nancey S, Buisson A, Pariente B, Fumery M, Sokol H, Treton X, Barnich N, Seksik P, Le Bourhis L; REMIND Study Group. T cell clonal expansions in ileal Crohn's disease are associated with smoking behaviour and postoperative recurrence. Gut. 2019 Nov;68(11):1961-1970. doi: 10.1136/gutjnl-2018-317878. Epub 2019 Feb 12. PMID 30792246
- [Result] Hammoudi N, Cazals-Hatem D, Auzolle C, Gardair C, Ngollo M, Bottois H, Nancey S, Pariente B, Buisson A, Treton X, Fumery M, Bezault M, Seksik P, Le Bourhis L; REMIND Study Group Investigators; Flejou JF, Allez M. Association Between Microscopic Lesions at Ileal Resection Margin and Recurrence After Surgery in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2020 Jan;18(1):141-149.e2. doi: 10.1016/j.cgh.2019.04.045. Epub 2019 Apr 28. PMID 31042575
- [Result] Fumery M, Seksik P, Auzolle C, Munoz-Bongrand N, Gornet JM, Boschetti G, Cotte E, Buisson A, Dubois A, Pariente B, Zerbib P, Chafai N, Stefanescu C, Panis Y, Marteau P, Pautrat K, Sabbagh C, Filippi J, Chevrier M, Houze P, Jouven X, Treton X, Allez M; REMIND study group investigators. Postoperative Complications after Ileocecal Resection in Crohn's Disease: A Prospective Study From the REMIND Group. Am J Gastroenterol. 2017 Feb;112(2):337-345. doi: 10.1038/ajg.2016.541. Epub 2016 Dec 13. PMID 27958285
- [Result] Khaloian S, Rath E, Hammoudi N, Gleisinger E, Blutke A, Giesbertz P, Berger E, Metwaly A, Waldschmitt N, Allez M, Haller D. Mitochondrial impairment drives intestinal stem cell transition into dysfunctional Paneth cells predicting Crohn's disease recurrence. Gut. 2020 Nov;69(11):1939-1951. doi: 10.1136/gutjnl-2019-319514. Epub 2020 Feb 28. PMID 32111634
- [Result] Perez K, Ngollo M, Rabinowitz K, Hammoudi N, Seksik P, Xavier RJ, Daly MJ, Dotan I, Le Bourhis L, Allez M. Meta-Analysis of IBD Gut Samples Gene Expression Identifies Specific Markers of Ileal and Colonic Diseases. Inflamm Bowel Dis. 2022 May 4;28(5):775-782. doi: 10.1093/ibd/izab311. PMID 34928348
- [Result] Ngollo M, Perez K, Hammoudi N, Gorelik Y, Delord M, Auzolle C, Bottois H, Cazals-Hatem D, Bezault M, Nancey S, Nachury M, Treton X, Fumery M, Buisson A, Barnich N, Seksik P; REMIND Study Group Investigators; Shen-Orr SS, Le Bourhis L, Allez M. Identification of Gene Expression Profiles Associated with an Increased Risk of Post-Operative Recurrence in Crohn's Disease. J Crohns Colitis. 2022 Aug 30;16(8):1269-1280. doi: 10.1093/ecco-jcc/jjac021. PMID 35143619
- [Result] Buisson A, Sokol H, Hammoudi N, Nancey S, Treton X, Nachury M, Fumery M, Hebuterne X, Rodrigues M, Hugot JP, Boschetti G, Stefanescu C, Wils P, Seksik P, Le Bourhis L, Bezault M, Sauvanet P, Pereira B, Allez M, Barnich N; Remind study group. Role of adherent and invasive Escherichia coli in Crohn's disease: lessons from the postoperative recurrence model. Gut. 2023 Jan;72(1):39-48. doi: 10.1136/gutjnl-2021-325971. Epub 2022 Mar 31. PMID 35361684
- [Result] Julien C, Anakok E, Treton X, Nachury M, Nancey S, Buisson A, Fumery M, Filippi J, Maggiori L, Panis Y, Zerbib P, Francois Y, Dubois A, Sabbagh C, Rahili A, Seksik P, Allez M, Lefevre JH; REMIND Study Group Investigators; Le Corff S, Bonnet A, Beyer-Berjot L, Sokol H. Impact of the Ileal Microbiota on Surgical Site Infections in Crohn's Disease: A Nationwide Prospective Cohort. J Crohns Colitis. 2022 Aug 30;16(8):1211-1221. doi: 10.1093/ecco-jcc/jjac026. PMID 35218661
- [Result] Chervy M, Sivignon A, Dambrine F, Buisson A, Sauvanet P, Godfraind C, Allez M, Le Bourhis L, The Remind Group, Barnich N, Denizot J. Epigenetic master regulators HDAC1 and HDAC5 control pathobiont Enterobacteria colonization in ileal mucosa of Crohn's disease patients. Gut Microbes. 2022 Jan-Dec;14(1):2127444. doi: 10.1080/19490976.2022.2127444. PMID 36175163
- [Result] Hammoudi N, Hamoudi S, Bonnereau J, Bottois H, Perez K, Bezault M, Hassid D, Chardiny V, Grand C, Gergaud B, Bonnet J, Chedouba L, Tran Minh ML, Gornet JM, Baudry C, Corte H, Maggiori L, Toubert A, McBride J, Brochier C, Neighbors M, Le Bourhis L, Allez M. Autologous organoid co-culture model reveals T cell-driven epithelial cell death in Crohn's Disease. Front Immunol. 2022 Nov 10;13:1008456. doi: 10.3389/fimmu.2022.1008456. eCollection 2022. PMID 36439157
- [Result] Hammoudi N, Auzolle C, Tran Minh ML, Boschetti G, Bezault M, Buisson A, Pariente B, Treton X, Seksik P, Fumery M, Le Bourhis L, Nancey S, Allez M. Postoperative Endoscopic Recurrence on the Neoterminal Ileum But Not on the Anastomosis Is Mainly Driving Long-Term Outcomes in Crohn's Disease. Am J Gastroenterol. 2020 Jul;115(7):1084-1093. doi: 10.14309/ajg.0000000000000638. PMID 32618659